CLINICAL TRIAL: NCT07123415
Title: A Phase 1 Trial of APX-343A as Monotherapy or in Combination With Pembrolizumab to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy in Subjects With Advanced Solid Tumors
Brief Title: A Phase 1 Study of APX-343A as Monotherapy or in Combination With Pembrolizumab in Subjects With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aptabio Therapeutics, Inc. (Individual)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APX-343A-101
Record Dates: First submitted 2025-07-29; First posted 2025-08-14 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Cancer; Advanced Solid Tumor (Phase 1)
Keywords: Advanced Solid Cancer; Advanced Solid Tumor (Phase 1); APX-343A; ICI; CAF; NOX
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A : APX-343A (Experimental): Part A is a dose-escalation study of APX-343A monotherapy in subjects with advanced solid tumors.
  Interventions: Drug: APX-343A
- Part B (Experimental): Part B is a dose-escalation study of APX-343A in combination with pembrolizumab, targeting subjects with advanced solid tumors.
  Interventions: Drug: APX-343A; Drug: Pembrolizumab

INTERVENTIONS:
Drug: APX-343A — Oral administration twice daily
Drug: Pembrolizumab — intravenous [IV]
  Arms: Part B

SUMMARY:
This is a Phase 1, open-label, dose-escalation study to assess the safety, tolerability, pharmacokinetics (PK), and preliminary efficacy of APX-343A monotherapy (Part A) and in combination with pembrolizumab (Part B) in subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥19 years, inclusive, at the time of informed consent.
2. Willing and able to give informed consent and to comply with the requirements of the study.
3. Histologically or cytologically confirmed advanced solid tumor.
4. Life expectancy of at least 3 months in the judgment of the investigator.
5. ECOG performance status of 0 to 1 during the screening period.
6. Measurable disease per RECIST v1.1 as assessed by the site investigator/radiology.
7. Archival tumor tissue sample or newly obtained biopsy of a tumor lesion not previously irradiated has been provided.
8. Subjects who have AEs due to previous anticancer therapies must have recovered to ≤ Grade 1 or baseline.
9. Adequate organ function as defined in the following table.
10. Subjects who are hepatitis B surface antigen positive are eligible if they have received HBV antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to the first dose of study drug.
11. Subjects with history of HCV infection are eligible if HCV viral load is undetectable at screening.
12. Male subjects must agree to use an adequate method of contraception.
13. Female subjects of childbearing potential must agree to use highly effective contraceptive methods, and to abstain from breastfeeding.

Exclusion Criteria:

1. Received any prior immunotherapy.
2. Received prior systemic anticancer therapy including investigational agents.
3. Received prior radiotherapy.
4. Received a live or live-attenuated vaccine .
5. Has received an investigational agent.
6. Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy.
7. Known additional malignancy.
8. Known active CNS metastases and/or carcinomatous meningitis.
9. Active autoimmune disease.
10. History of (noninfectious) pneumonitis/interstitial lung disease.
11. Active, uncontrolled infection requiring systemic therapy.
12. Unable to swallow study drug or disease that interfere with proper absorption of study drug.
13. Significant cardiovascular disease.
14. Cerebrovascular accident.
15. History or current evidence of any condition, therapy, laboratory abnormality, or other circumstance that might confound the results of the study or interfere with the subject's ability to cooperate with the requirements of the study.
16. History of severe hypersensitivity to pembrolizumab and/or any of its excipients.
17. History of hypersensitivity to APX-343A and/or any of its excipients.
18. History of allogeneic tissue/solid organ transplant.
19. History of HIV infection or HIV positive at screening.
20. Subjects who have not adequately recovered from major surgery or have ongoing surgical complications.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability and to determine the MTD and/or RP2D of APX-343A monotherapy and in combination with pembrolizumab | From enrollment to 90 days after End Of Treatment
  Number and severity of TEAEs according to NCI-CTCAE v5.0

SECONDARY OUTCOMES:
Cmax of APX-343A | From enrollment to 3 weeks
  To characterize the PK of APX 343A monotherapy
AUC of APX-343A | From enrollment to 3 weeks
  To characterize the PK of APX-343A monotherapy
Tmax of APX-343A | From enrollment to 3 weeks
  To characterize the PK of APX-343A monotherapy
t1/2 of APX-343A | From enrollment to 3 weeks
  To characterize the PK of APX-343A monotherapy
CL of APX-343A | From enrollment to 3 weeks
  To characterize the PK of APX-343A monotherapy
Response rate according to RECIST v1.1 and iRECIST | Through study completion, an average of 1 year
  To evaluate preliminary efficacy of APX-343A monotherapy and in combination with pembrolizumab

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul